CLINICAL TRIAL: NCT02399475
Title: The Thyroid Axis in Older Individuals With Persistent Subclinical Hypothyroidism: a Mechanistic, Randomized, Double-Blind, Cross-Over Study of Levothyroxine and Liothyronine Administration
Brief Title: Mechanistic Study of Subclinical Hypothyroidism In the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 821564; K24AG042765-01A1 (NIH)
Record Dates: First submitted 2015-02-03; First posted 2015-03-26 (Estimated); Results first posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-02

CONDITIONS: Subclinical Hypothyroidism
Keywords: Levothyroxine; Liothyronine; Thyrotropin Releasing Hormone; Aging; Hypothyroidism; Thyroid diseases
MeSH Terms: conditions — Hypothyroidism; Thyroid Diseases | interventions — Thyroxine; Triiodothyronine; Thyrotropin-Releasing Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levothyroxine First (Experimental): Participants will start on the thyroid hormone Levothyroxine prior to crossing over to Liothyronine
  Interventions: Drug: Levothyroxine; Drug: Liothyronine; Drug: Thyrotropin-Releasing Hormone
- Liothyronine First (Experimental): Participants will start on the thyroid hormone Liothyronine prior to crossing over to Levothyroxine
  Interventions: Drug: Levothyroxine; Drug: Liothyronine; Drug: Thyrotropin-Releasing Hormone

INTERVENTIONS:
Drug: Levothyroxine — Oral levothyroxine with a total starting dose of 0.7mcg/kg/day split into three daily doses will be titrated to a target TSH level of 0.5 -1.5mU/L
  Other Names: Synthroid
Drug: Liothyronine — Oral liothyronine with a starting dose of 1/3 of the weight-based LT4 dose divided into three daily doses titrated to a target TSH level of 0.5 -1.5mU/L
  Other Names: Cytomel
Drug: Thyrotropin-Releasing Hormone — 200 µg intravenous TRH will be given at study visit 1 (baseline), study visit 2 (on first thyroid treatment), and study visit 3 (on second thyroid treatment).

SUMMARY:
Subclinical hypothyroidism, defined as an elevated TSH in the setting of normal thyroid hormone levels, is a common diagnosis in the elderly. The purpose of this study is to examine the hypothalamic-pituitary-thyroid axis in men and women aged 70 years and older with persistent subclinical hypothyroidism. To evaluate the mechanism behind this condition, participants will undergo thyrotropin releasing hormone stimulation testing at 3 visits: baseline and while taking two different thyroid hormone preparations, levothyroxine and liothyronine. The investigators will also assess physiologic responses to these two different thyroid hormone medications to help us understand how the thyroid works in advanced age.

ELIGIBILITY:
Inclusion Criteria:

1. men and women aged 70 and older
2. TSH between 4.5 and 19.9 mU/L as an outpatient
3. ability to provide informed consent

Exclusion Criteria:

Laboratory Tests:

1. TSH <4.5 mU/L or >20 mU/L on repeat testing at least four weeks later or free T4 level outside the reference range
2. thyroid peroxidase (TPO) antibody positive
3. abnormal liver function tests (LFTs >3 x upper limit of normal)
4. hemoglobin <11 g/dL

Surgeries or Procedures:

1. thyroid surgery
2. pituitary surgery
3. bariatric surgery
4. bowel resection involving the jejunum and upper ileum
5. radioactive iodine therapy
6. radiation treatments to head or neck

Medical Conditions:

1. diagnosis of pituitary disease
2. diagnosis of amyloidosis, sarcoidosis, hemochromatosis
3. diagnosis of adrenal insufficiency
4. obesity with BMI > 35 mg/kg2
5. history of stroke
6. chronic or ongoing angina, Class II or higher congestive heart failure, or uncontrolled hypertension with current blood pressure greater than 160/100
7. diabetes mellitus with hemoglobin A1C level greater than 8.0% in the past six months
8. celiac sprue, Crohn's disease, ulcerative colitis, Zollinger-Ellison syndrome
9. renal insufficiency with calculated glomerular filtration rate <45 cc/min
10. cognitive impairment with Mini Mental State Exam[30] <24/30
11. history of any seizures
12. unstable medical or psychological condition in the judgment of the principal investigator

Medications:

1. thyroid hormone preparations
2. antithyroid drugs
3. medications that interfere with the absorption or metabolism of thyroid hormone
4. medications that interfere with the TRH stimulation test
5. proton pump inhibitors

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne R Cappola, MD, ScM, Principal Investigator — The University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Levothyroxine First | Liothyronine First
Started | 7 | 7
Completed | 6 | 7
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levothyroxine First | Liothyronine First | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 77 (5) | 77 (4) | 77 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 4 | 5 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 7 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: TSH Area Under the Curve
Description: TSH area under the curve within 60 minutes of TRH stimulation when TSH is at goal
Time Frame: 0, 5, 10, 15, 20, 30, and 60 min post TRH
Measure: Mean (Standard Deviation); unit: μIU*min/mL
Groups:
- Levothyroxine: While taking levothyroxine
- Liothyronine: While taking liothyronine
Arm/Group | Levothyroxine | Liothyronine
Number analyzed (Participants) | 13 | 13
μIU*min/mL | 267.8 (137.3) | 266.2 (140.2)

2. Primary Outcome: TSH Max
Description: The maximum concentration of TSH after TRH stimulation when TSH is at goal
Time Frame: Between 0 and 180 min after TRH stimulation
Measure: Mean (Standard Deviation); unit: mIU/L
Arm/Group | Levothyroxine | Liothyronine
Number analyzed (Participants) | 13 | 13
mIU/L | 5.5 (3.0) | 5.4 (2.9)

3. Primary Outcome: Free T4 Level
Description: Free thyroxine level when TSH level is at goal on therapy.
Time Frame: An average of 7 months after initiating therapy
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Levothyroxine | Liothyronine
Number analyzed (Participants) | 13 | 13
ng/dL | 1.65 (0.11) | 0.46 (0.19)

4. Primary Outcome: Total T3 Level
Description: Total triiodothyronine level when TSH is at goal on therapy
Time Frame: An average of 7 months
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Levothyroxine | Liothyronine
Number analyzed (Participants) | 13 | 13
ng/mL | 1.12 (0.24) | 1.98 (0.51)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 7 months in each arm
Arm/Group | Levothyroxine | Liothyronine
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/75/NCT02399475/Prot_SAP_000.pdf